CLINICAL TRIAL: NCT03356327
Title: Oral Administration of Tannins and Flavonoids in Children With Acute Diarrhea : A Pilot, Randomized, Control-case Study
Brief Title: Oral Administration of Tannins and Flavonoids in Children With Acute Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Annamaria Staiano, Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/11/2017
Record Dates: First submitted 2017-11-16; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Acute Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 consisting of 30 children treated with Actitan F and standard oral rehydration (SOR)
  Interventions: Drug: Actitan F; Drug: Standard Oral Rehydration
- Group 2 (Active Comparator): Group 2 consisting of 30 children who received only SOR.
  Interventions: Drug: Standard Oral Rehydration

INTERVENTIONS:
Drug: Actitan F — A molecolar complex of Tannins and Flavonoids used for acute diarrhea in children
  Arms: Group 1
Drug: Standard Oral Rehydration — Standard oral rehydration as suggested by ESPGHAN guidelines

SUMMARY:
A pilot, randomized, case-controlled trial was conducted in 60 children affected by AG (< 7 days) with mild-moderate dehydration, according to WHO recommendations, from1 year to 17 years old. Patients were divided into 2 Groups: Group 1 consisting of 30 children treated with Actitan F and standard oral rehydration (SOR); Group 2 consisting of 30 children who received only SOR. Both groups received treatment for seven days, respectively. Patients of Group 1 stopped for their own choice, SOR after the first 24 h and continued only with Actitan F.

DETAILED DESCRIPTION:
The investigators included 60 children (mean age: 3.1yrs, range 0.3-12years) with a diagnosis of AG, referred between April and July 2017 to the Department of Translational Medicine, section of Pediatric, University of Naples Federico II.

Patients enrolled were children from 3 months to 12 years old, with a diagnosis of acute diarrhea appeared less than 7 days before the admission, capability to oral rehydration, mild to moderate dehydration. Patients with diarrhea over 7 days, serious somatic pathology and severe dehydration were excluded.

The study was approved by the Institutional Review Board of the University of Naples "Federico II" with the protocol number 25/17. At admission, written informed consent was obtained from participants' parents and from all patients older than 10 years. At first visit, a medical history was collected by one of the authors and all patients underwent clinical evaluation, including body weight and body temperature.

Frequency of bowel movements, stool consistency measured through the Bristol Stool Form Scale (BSFS) and other associated gastrointestinal symptoms, including nausea, vomiting, abdominal pain and rectal bleeding, were accurately recorded. The BSFS is the most commonly standardized instrument used to rate stool consistency in children. On admission, the degree of dehydration was clinically determined for each patient, based on WHO recommendations and data were recorded on a scale from 1 to 3 (1 for mild or <5%; 2 for moderate or 5% to 10%; 3 for severe or 10% and more).

Participants were randomly divided into two groups: Group 1 was treated with Actitan F and standard oral rehydration (SOR) and Group 2 was treated with SOR only ad libitum for 7 days. SOR is a reduced osmolarity oral solution (50/60 mmol/L Na), which is the first line therapy recommended by ESPGHAN guideline for Acute Diarrhea. Actitan F, instead, was orally administrated at dose of 1 sack every 4 hours, maximum 4 sacks/day for 7 days. Caregivers were instructed to administer the daily dose after mixing the contents of the sachet with a small amount of water. The study products used in this trial were donated by Aboca® Società Agricola SpA., Località Aboca, 20, 52037 Sansepolcro (AR) - Italy.

At home, all parents had to fulfill a daily diary to record number and consistency of stools, presence of fever, vomiting and children compliance with the therapy. During the final visit, scheduled after 7 days, the interim history was assessed, daily diaries were reviewed and discussed, and a physical evaluation was performed.

Outcomes

The primary outcome was the duration of diarrhea, defined as the number of stools after 24 hours of treatment or the time needed to normalize number and consistency of stools (compared with the period before the onset of diarrhea). Secondary outcomes were the evaluation of vomiting, body weight, possible need of hospitalization, compliance to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled were children from 3 months to 12 years old, with a diagnosis of acute diarrhea appeared less than 7 days before the admission, capability to oral rehydration, mild to moderate dehydration.

Exclusion Criteria:

* Patients with diarrhea over 7 days, serious somatic pathology and severe dehydration were excluded.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
effectiveness of a medical device made of Actitan-F in the treatment of acute diarrhea, valuated on the basis of consistency of stools based on Bristol Stool Form | 2 weeks
  the effectiveness of a medical device made of Actitan-F, a natural molecular complex of tannins (from Agrimony and Tormentil) and flavonoids (Chamomile), in the treatment of acute gastroenteritis (AG) in children, valuated on the basis of stool consistency
effectiveness of a medical device made of Actitan-F in the treatment of acute diarrhea, valuated on the basis of number of stools / day | 2 weeks
  he effectiveness of a medical device made of Actitan-F, a natural molecular complex of tannins (from Agrimony and Tormentil) and flavonoids (Chamomile), in the treatment of acute gastroenteritis (AG) in children, valuated on the basis of number of stools/day

CONTACTS AND LOCATIONS:
Locations (1):
- Marina Russo, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russo M, Coppola V, Giannetti E, Buonavolonta R, Piscitelli A, Staiano A. Oral administration of tannins and flavonoids in children with acute diarrhea: a pilot, randomized, control-case study. Ital J Pediatr. 2018 Jun 4;44(1):64. doi: 10.1186/s13052-018-0497-6. PMID 29866147